CLINICAL TRIAL: NCT02376582
Title: A Phase I Double Blind Placebo-controlled Clinical Trial to Evaluate the Safety and Immunogenicity of the Combination of DNA-HIV-PT123 and AIDSVAX®B/Ein HIV-1-uninfected Adult Participants With or Without Underlying Schistosoma Mansoni Infection
Brief Title: Safety and Immunogenicity Study of a DNA Vaccine Combined With Protein Vaccine Against HIV/AIDS
Acronym: EV06
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EuroVacc Foundation (Other)
Collaborators: International AIDS Vaccine Initiative (Network); Medical Research Council (Other Government); MRC/UVRI and LSHTM Uganda Research Unit (Other); Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EV06
Record Dates: First submitted 2014-07-18; First posted 2015-03-03 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS vaccine; helminth infection; Impact of co-infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Trematode Infections | interventions — DNA; AIDSVAX B-E

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DNA and protein (Experimental): 4mg DNA and 600 mcg protein formulated with Alum co-administration (IM) at Month 0, 1 and 6 in Schisto infected individuals
  Interventions: Biological: DNA; Biological: AIDSVAX B/E
- Vaccination without S. mansoni infection (Active Comparator): DNA Protein
  Interventions: Biological: DNA; Biological: AIDSVAX B/E

INTERVENTIONS:
Biological: DNA — DNA co-administered with protein at month 0, 1 and 6
  Other Names: DNA-HIV-PT123
Biological: AIDSVAX B/E — Protein co-administered with DNA at month 0,1 and 6

SUMMARY:
The primary objective of the proposed phase I trial is to evaluate the safety and tolerability of DNA-HIV-PT123 and AIDSVAX®B/E combination regimen. Though both DNA-HIV-PT123 and AIDSVAX®B/E and the combination of the two vaccines have been evaluated in humans and have shown to be safe and well tolerated, this is the first time the combination regimen is being evaluated in HIV-1 uninfected African populations with and without S. mansoni. The secondary objective of the trial is to evaluate the effect of S. mansoni infection on the immunogenicity of the combination of DNA-HIV-PT123 and AIDSVAX® B/E vaccine regimen. Successful vaccination against most viruses requires efficient Th1 response. There is evidence that helminth infections skew the host immune system of human and animals to T-helper type 2 (Th2) and induce immunosuppression. Therefore, there is a potential that helminth infected populations may not generate the desired immune responses to vaccines designed to drive Th1-type and cytotoxic T-cell responses.

Furthermore, the influence of helminth infections on the development of protective antibody responses remains unclear. Limited data in animal models suggests that worm infections reduced efficacy of vaccines.

The proposed vaccine trial will generate safety, tolerability and immunogenicity data of a vaccination regimen with simultaneous administration of a candidate HIV DNA vaccine (DNA-HIV-PT123) and a gp120 protein vaccine (AIDSVAX®B/E). This will be the first HIV vaccine trial to prospectively evaluate the impact of the S. mansoni infection on safety and immune responses to HIV vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 uninfected adults aged 18-45 years, as confirmed by a medical history, physical exam, and laboratory tests during screening
2. In 50% of study volunteers, positive for S. mansoni infection but negative for other helminth infections.
3. In 50% of study volunteers, negative for S. mansoni and other helminth infections
4. Willing to forgo treatment with praziquantel until after completion of week 26 visit in the trial.
5. Able and willing to provide written informed consent prior to screening
6. Aged 18 through 45 years on the day of first vaccination
7. Able and willing to complete screening (about 1 month) and available for the planned follow-up period (9months)
8. Willing to undergo HIV testing, risk reduction counselling, receive HIV test results and committed to maintaining low risk behaviour for the trial duration
9. If female of childbearing potential (not menopausal or sterilised), willing to use a non-barrier contraceptive method from screening through the end of the study. Acceptable contraceptive methods include hormonal contraceptives (injection, transdermal patch, or implant) and intrauterine device (IUD).
10. Willing to provide blood, urine and stool samples for laboratory examination

Exclusion Criteria:

1. HIV-1 infection
2. Infection with other helminths
3. Symptomatic and asymptomatic malaria infection (presence of malaria parasites on thick blood smear)
4. Treatment with praziquantel in the past 3 months
5. S. mansoni egg count of>2000 eggs per gram of stool
6. Clinically significant acute or chronic illness at the time of randomization.
7. Any clinically relevant abnormality on history or examination
8. Use of immunosuppressive medication (other than inhaled or topical immunosuppressants)
9. Receipt of immunoglobulin within past 60 days
10. Abnormal laboratory values as specified below from blood collected within 28 days prior to randomization:

    1. Hematology

       * Haemoglobin <9.0 g/dL or<5.59 mmol/L
       * Absolute Neutrophil Count (ANC): < 1000/mm3or < 1.0 x 109/L
       * Absolute Lymphocyte Count (ALC): ≤ 500/mm3or ≤ 0.5 x 109/L
       * Platelets: ≤ 90,000 ≥ 550,000/mm3or ≤ 90 x 109 ≥ 550 x 109/L
    2. Chemistry

       * Creatinine: > 1. 1 x ULN
       * AST: >2.6 x ULN
       * ALT: >2.6 x ULN
    3. Urinalysis: abnormal dipstick confirmed by microscopy

       * Protein 2+ or more
       * Blood 2+ or more (not due to menses)
11. Reported high-risk behaviour for HIV infection within 3 months prior to first vaccination, as defined by:

    * Unprotected sexual intercourse with a known HIV-infected person, a partner known to be at high risk of HIV infection or a casual partner
    * Unprotected sexual intercourse with more than one sexual partner
    * Engagement in sex work for money or drugs
    * Use of recreational drugs (e.g. marijuana) and/or weekly or more frequent alcohol use
    * Current or past STI
12. History or evidence of autoimmune disease.
13. Positive for Hepatitis B surface antigen (HbsAg), positive for antibodies to Hepatitis C virus (HCV) or active syphilis.
14. Receipt of blood or blood products within the previous 6 months
15. History of severe allergic reactions to any substance requiring hospitalization or emergency medical care (e.g. Steven-Johnson syndrome, bronchospasm or hypotension)
16. Prior or current participation in another investigational agent trial
17. Current anti-tuberculosis (TB) prophylaxis or therapy
18. If female, currently pregnant (positive serum or urine pregnancy test), planning to get pregnant in the next 9months or lactating
19. History or evidence of any systemic disease or any acute or chronic illness that, in the opinion of the investigator, may compromise the volunteer's safety or interfere with the evaluation of the safety or immunogenicity of the vaccine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2014-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Proportion of volunteers with local and systemic reactogenicity events during a 7 day follow up period after each vaccination | 7 days post each vaccination
Proportion of volunteers with adverse events during a 4 week follow up period after each vaccination | 4 weeks post each vaccination
Proportion of volunteers with abnormal laboratory parameters during a 4 week follow up period after each vaccination | 4 weeks post each vaccination
Proportion of volunteers with serious adverse events throughout the study period | Each participant will be followed for 9 months

SECONDARY OUTCOMES:
Proportion of volunteers with HIV-specific CD4+ and CD8+ T cell responses as assessed by IFN-g ELISpot and multiparameter flow cytometry (IFN-g TNF-a and IL-2) 2 weeks after the 2nd and 3rd vaccination | two weeks post 2nd and 3 vaccination
Magnitude of HIV-specific CD4+ and CD8+ T cell responses as assessed by IFN-g ELISpot and multiparameter flow cytometry (IFN-g TNF-a and IL-2) 2 weeks after the 2nd and 3rd vaccination | two weeks post 2nd and 3 vaccination
HIV-specific Env binding Antibody response 2 weeks after the 2nd and 3rd vaccination | two weeks post 2nd and 3 vaccination
Magnitude and breadth of neutralizing antibody responses against tier 1 and tier 2 HIV-1 isolates 2 weeks after the 2nd and 3rd vaccination | two weeks post 2nd and 3 vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Pontiano Kaleebu, Principal Investigator — Medical Research Council (MRC) / Uganda Virus Research Institute (UVRI)
Locations (2):
- Uganda (2):
  - Uganda Virus Research Institute - International AIDS Vaccine Initiative HIV Vaccine Program (UVRI-IAVI), Entebbe
  - Medical Research Council (MRC) /Uganda Virus Research Institute (UVRI), Masaka